CLINICAL TRIAL: NCT04208815
Title: Evaluation of Dietary Milk Polar Lipids on Serum Cholesterol and Gut Microbiota in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Christopher Blesso, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H19-122
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Serum Cholesterol; Gut Microbiome
Keywords: Milk; Polar Lipids; Phospholipids; Cholesterol; Microbiota; Microbiome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPL-rich dairy beverage (Experimental): Daily consumption of 100 g of dairy powder containing 5.3 g MPL for 4 weeks
  Interventions: Other: Milk Polar Lipids; Other: Milk Fat
- Control dairy beverage (Placebo Comparator): Daily consumption of 100 g of dairy powder containing 0.3 g MPL for 4 weeks
  Interventions: Other: Milk Fat

INTERVENTIONS:
Other: Milk Polar Lipids — Effects of the addition of 5 g of milk polar lipids to 20 g milk fat.
  Arms: MPL-rich dairy beverage
Other: Milk Fat — Effects of the addition of 20 g milk fat.

SUMMARY:
The purpose of this study is to examine whether the daily consumption of 5 g of milk polar lipids influences serum lipids and gut microbiota composition in healthy adults.

DETAILED DESCRIPTION:
Healthy adults will be recruited to participate in a randomized, single-blind, controlled, 13-week crossover trial. Participants will follow a 2-week run-in control period consuming their habitual diets. Participants will then be randomized to consume 20 g of milk fat daily in the form of either a reconstituted milk polar lipid (MPL)-rich dairy beverage (MPL; providing 5.3 g MPL daily) or a control dairy beverage (CTL; providing 0.3 g MPL daily), each for 4- weeks, separated by a 3-week washout period. Participants will be instructed to consume intervention treatment/control beverages at breakfast (50 g) and dinner (50 g) and reconstitute the powders in water immediately prior to consumption. With the exception of the intervention beverages, participants will be asked to maintain their normal diet and exercise habits throughout the study. Venous blood will be collected after a 12-hour overnight fast into EDTA-coated (glucose analysis) and serum (lipid analyses) collection tubes. Passive drool and stool samples will be collected at the end of the run-in period (baseline) and intervention periods (treatment and control). Participants will be asked to complete a 5-day dietary record, food preference/liking/sedentary behavior surveys, and 7-day physical activity diary at the beginning and end of intervention periods.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 50 years
* Body Mass Index < 30 kg/m^2
* Willing to consume experimental intervention products on a daily basis

Exclusion Criteria:

* Outside of age range (<18 or >50 years old)
* Body Mass Index > 30 kg/m^2
* Triglycerides are higher than 500 mg/dL, glucose levels higher than 126 mg/dL, or total cholesterol higher than 240 mg/dL
* Self-reported history of renal or liver disease, diabetes, thyroid disease, gallbladder disease, eating disorders, heart disease, stroke, cancer and gut-associated pathologies
* Weight loss greater than 10% of body weight over preceding 4 weeks
* Taking probiotic supplements or oral antibiotics up to 1 month prior to the study and during the study
* Allergy to dairy or lactose intolerance
* Taking lipid-lowering medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Serum Total Cholesterol at 4 weeks | 4 weeks
  Measurement of serum cholesterol (mg/dL) at the beginning and end of each 4-week intervention arms.

SECONDARY OUTCOMES:
Change in Fecal Microbiota Shannon Index at 4 weeks | 4 weeks
  Measurement of fecal microbiota Shannon Index at the end of each 4-week intervention arms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States